CLINICAL TRIAL: NCT02551029
Title: Brain and Brainstem Activation Following Duodenal Nociceptive Stimulation With Capsaicin, an Exploratory High-resolution fMRI Study in Healthy Volunteers
Brief Title: fMRI and Visceral Perception Upon Capsaicin Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 152048; NL51770.068.15 (Other: CCMO); METC 152048 (Other: METC Azm/UM)
Record Dates: First submitted 2015-08-25; First posted 2015-09-16 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Irritable Bowel Syndrome; Colonic Diseases, Functional; Dyspepsia; Gastrointestinal Diseases; Abdominal Pain; Visceral Pain
Keywords: Magnetic Resonance Imaging; Brainstem; Solitary Nucleus; Visceral Nervous System; Transient Receptor Potential Channels
MeSH Terms: conditions — Irritable Bowel Syndrome; Colonic Diseases, Functional; Dyspepsia; Gastrointestinal Diseases; Abdominal Pain; Visceral Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duodenal capsaicin infusion (Experimental): Through a naso-duodenal tube, a capsaicin solution will be infused into the duodenum.
  Interventions: Other: Capsaicin
- Placebo (saline) (Placebo Comparator): Through a naso-duodenal tube, a saline solution will be infused into the duodenum.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Capsaicin
  Other Names: Capsaicin oleoresina solution infusion into the duodenum.
  Arms: Duodenal capsaicin infusion
Other: Placebo
  Other Names: Saline infusion into the duodenum
  Arms: Placebo (saline)

SUMMARY:
Brain imaging has shown abnormal brain activations in response to visceral stimulation in patients with the Irritable Bowel Syndrome (IBS) and Functional Dyspepsia (FD). To investigate the possible role of the Nucleus of the Solitary Tract (NTS), the primary relay station in the brainstem for vagal afferents, its activation in IBS and functional dyspepsia patients will be evaluated. Prior to this, an exploratory study in healthy volunteers will be conducted. This will be the first high magnetic field fMRI study (7T) evaluating the possible role of NTS activation in visceral abdominal pain. Moreover, this will be the first pharmacological fMRI study using duodenal capsaicin infusion as a chemical stimulus, which is more physiological than mechano-stimulation in the upper gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Of female sex
* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years.
* BMI between 18 and 30 kg/m2
* Women in fertile age (<55 years old) must use contraception or be postmenopausal for at least two years.
* All subjects should be right-handed.

Exclusion Criteria:

* Presence of metallic prostheses, pacemakers, metal clips on blood vessels, metal parts in the eye, an intrauterine device, metal braces, tattoos and/or other metal objects;
* History of major head trauma or head/brain surgery;
* History of claustrophobia;
* History of severe or chronic cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol;
* Use of medication, including vitamin and iron supplementation, except oral contraceptives, within 14 days prior to start of the study;
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgment of the principle investigator);
* Pregnancy, lactation, wish to become pregnant;
* High alcohol consumption (>15 alcoholic consumptions per week);
* Using drugs of abuse;
* Self-admitted HIV-positive state;
* Known allergic reaction to capsaicin;
* High intake of spicy (capsaicin containing) food (meaning an estimated intake of > than 1.5mg/day), due to possible desensitization of the capsaicin receptor TRPV1 (see further below);
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study;
* Any evidence of structural brain abnormalities examined by anatomical MRI will lead to exclusion.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Activation of the Nucleus of the Solitary Tract | During duodenal capsaicin and placebo infusion between t=0 and and t=38 minutes
  the BOLD (Voxel-wise blood oxygenation level dependent) signal activity in the Nucleus of the Solitary Tract during capsaicin infusion compared to placebo

SECONDARY OUTCOMES:
Activity and connectivity in the Cingulate Cortex, Insula, Thalamus, Prefrontal Cortex, Primary and Secondary Somatosensory Cortex, Amygdala, PAG | During duodenal capsaicin and placebo infusion between t=0 and and t=60 minutes
  the functional BOLD signal activity in the above-mentioned brain structures during capsaicin infusion compared to placebo
Questionnaire for pain (Visual Analogue Scores) | During capsaicin and placebo infusion between t=0 and and t=38 minutes
  Scores range from 0 [no pain] to 10 [worst possible pain].
Questionnaire for depression and anxiety | During the test day, before scanning
  Hospital Anxiety and Depression Scale (HADS). Has 14 items (7 for depression, 7 for anxiety) with a 4 points likert scale (0-3). Scores for depression and anxiety range from 0-21 and studies identified 8 as the cutoff-point.
Questionnaire for depression | During the test day (= day 1), before scanning
  PHQ-9 scores (patient health questionnaire). The questionnaire has 9 items with a 4 points likert scale (0-3) and a total score of 27. A total score of 0-4 indicates none to minimal depressive symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Questionnaire for personality trait | During the test day (= day 1), before scanning
  BIG FIVE Inventory, the Big Five Inventory (BFI) survey that measures the big five dimensions of personality (extraversion, neuroticism, consciousness, agreeableness, and openness to experience). The questionnaire has 44 items.
Questionnaire for quality of life | During the test day (= day 1), before scanning
  SF-36 (quality of life) scores, The Short Form (36) Health Survey questionnaire of 36 items, scale 1-6, generates a physical and a mental QoL component summary.
Questionnaire for current affect scores | During the test day (= day 1), before scanning
  PANAS-SF (current affect) scores, Positive and Negative Affect Schedule. This is a 20 item questionnaire (scale 1-5) total scores can range from 10 - 50, with higher scores representing higher levels of positive affect.
Questionnaire for current pain | During the test day (= day 1), before scanning
  Brief Pain Inventory (BPI) scores, The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub- items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Questionnaire for anxiety | During the test day (= day 1), before scanning
  GAD-7 scores, for screening and severity measuring of generalized anxiety disorder (GAD). GAD-7 has seven items, 0-3 scale.
Questionnaire for the assessment of Gastrointestinal symptom scores | During the test day (= day 1), before scanning
  Scores of the GSRS, scale 1-7, generates subscores for abdominal pain, reflux, diarrhea, constipation, indigestion
Questionnaire for the assessment of Gastrointestinal symptom scores | During the test day (= day 1), before scanning
  Scores of the GSRS-IBS, scale 1-7, generates subscores for abdominal pain, bloating, constipation, diarrhea, satiety.
Questionnaire for the assessment of early life traumata | During the test day (= day 1), before scanning
  Scores of the ETISR-SF, The Early Trauma Inventory Self Report - Short Form comprises of 27 items, divided into four dimensions (general trauma, physical abuse, emotional abuse and sexual abuse) and scored on a dichotomous scale (Yes/No).
Questionnaire for the assessment of gastrointestinal specific anxiety | During the test day (= day 1), before scanning
  Scores of the Visceral Sensitivity Index, a 15 item questionnaire, scale 1-6, assesses gastrointestinal (GI)-specific anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Prof. MD. PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Beckers AB, van Oudenhove L, Weerts ZZRM, Jacobs HIL, Priovoulos N, Poser BA, Ivanov D, Gholamrezaei A, Aziz Q, Elsenbruch S, Masclee AAM, Keszthelyi D. Evidence for engagement of the nucleus of the solitary tract in processing intestinal chemonociceptive input irrespective of conscious pain response in healthy humans. Pain. 2022 Aug 1;163(8):1520-1529. doi: 10.1097/j.pain.0000000000002538. Epub 2021 Nov 15. PMID 34799534